CLINICAL TRIAL: NCT04829435
Title: A Phase I Randomized, Double-Blind, Placebo Controlled, Multiple Ascending Dose Study of ALLN-346 (Engineered Urate Oxidase)
Brief Title: Study 102: Multiple Ascending Dose Study of ALLN-346 (Engineered Urate Oxidase)
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLN-346-102
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-03

CONDITIONS: Hyperuricemia; Gout
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLN-346 (Engineered Urate Oxidase) (Experimental): ALLN-346 is novel urate oxidase provided as capsules for oral administration. Two ascending dose cohorts: Cohort A (3 capsules thrice daily (TID) for a total of 9 capsules per day) and Cohort B (5 capsules thrice daily (TID) for a total of 15 capsules per day) will be evaluated for 7 days for each cohort.
  Interventions: Drug: ALLN-346
- Placebo (Placebo Comparator): Matching placebo capsules for oral administration. Two ascending dose cohorts: Cohort A (3 capsules thrice daily (TID) for a total of 9 capsules per day) and Cohort B (5 capsules thrice daily (TID) for a total of 15 capsules per day) will be evaluated for 7 days for each cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALLN-346 — ALLN-346 (Engineered Urate Oxidase) is an orally administered, novel urate oxidase; provided as capsules for oral administration; It is a proprietary enzyme designed to degrade urate in the intestinal tract
  Other Names: Engineered urate oxidase
  Arms: ALLN-346 (Engineered Urate Oxidase)
Drug: Placebo — Matched placebo capsules are similar in weight and appearance to the ALLN-346 capsules
  Other Names: Matching placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this Phase I study is to evaluate the safety and tolerability of ALLN-346 in in normal healthy volunteers, in an ascending dose design.

ALLN-346 is an (oral) enzyme that specifically degrades urate in the intestinal tract.

DETAILED DESCRIPTION:
This is a Phase I, 7-day, randomized, double-blind, placebo-controlled, multiple ascending dose study of orally administered ALLN-346 in normal healthy volunteers. Study will take place at a clinical pharmacology unit (CPU). Two sequential cohorts will be dosed and followed for safety through Day 28.

The study will evaluate safety and tolerability (including inflammation and immunogenicity), and pharmacodynamics of ALLN-346.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 55 years
* Incapable of pregnancy, not nursing, and agrees to use an effective method of contraception; males subjects must agree to abstain from sperm donation
* Good general health as determined by medical history and physical examination
* Normal clinical laboratory test results and ECG

Exclusion Criteria:

* Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurological, psychiatric disease or history of hyperuricemia
* Any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines
* Positive screen results for drugs of abuse, alcohol, or cotinine or recent history of drug or alcohol abuse, or positive COVID-19 test
* Clinically significant abnormal findings on physical examination, vital signs or on electrocardiogram (ECG)
* Positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody
* Received treatment with or exposure to an Investigational drug or device within 30 days prior to or during Screening
* Prior dosing in ALLN-346 clinical study
* Per Investigator judgment, is not an ideal clinical study candidate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 28 days
  Number of of participants with treatment emergent adverse events

SECONDARY OUTCOMES:
Serum ALLN-346 | 8 days
  Change of serum concentration of ALLN-346 (ng/mL) and uricase activity (mU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Tosone, MS, RAC, Study Director — Allena Pharmaceuticals, Inc.
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No